CLINICAL TRIAL: NCT04241315
Title: A Phase 3, Randomized,Single Dose, Open-Label Study to Investigate the Safety and Efficacy of OTL38 Injection for Intraoperative Imaging of Folate Receptor Positive Lung Nodules
Brief Title: ELUCIDATE: Enabling Lung Cancer Identification Using Folate Receptor Targeting
Acronym: Elucidate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: On Target Laboratories, LLC (Industry)
Collaborators: Clinipace Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OTL-2019-OTL38-007
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-01

CONDITIONS: Lung Neoplasms; Lung Cancer
Keywords: Intraoperative Imaging
MeSH Terms: conditions — Lung Neoplasms | interventions — Pafolacianine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Near-Infrared Imaging group (Experimental): All patients in this arm will receive OTL38 for injection and undergo intraoperative imaging.
  Interventions: Drug: OTL38 for Injection; Device: Near infrared camera imaging system
- No Imaging Group (Other): All patients in this arm will receive OTL38 for injection but will not receive intraoperative imaging.
  Interventions: Drug: OTL38 for Injection

INTERVENTIONS:
Drug: OTL38 for Injection — Folate analog ligand conjugated with an indole cyanine-like green dye as a solution in vials containing 3 mL at 2 mg/mL
  Other Names: CYTALUX™ (pafolacianine) injection
Device: Near infrared camera imaging system — Near infrared camera imaging system
  Arms: Near-Infrared Imaging group

SUMMARY:
This is a phase 3, multi-center, single dose, open-label, exploratory study in suspected lung cancer patients scheduled to undergo endoscopic or thoracic surgery per CT/PET/MRI or other imaging based on standard of care. This study aims to assess the efficacy of OTL38 and Near Infrared Imaging (NIR) at identifying pulmonary nodules within the operating theater, and to assess the safety and tolerability of single intravenous doses of OTL38.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female subjects 18 years of age and older
2. Have a primary diagnosis, or a high clinical suspicion, of cancer in the lung warranting surgery based on CT/PET or other imaging
3. Are scheduled to undergo surgical thoracoscopy for diagnostic wedge resection followed by anatomic lung resection
4. Female subjects of childbearing potential or less than 2 years postmenopausal agree to use an acceptable form of contraception from the time of signing informed consent until 30 days after study completion
5. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for the required assessments

Exclusion Criteria:

1. Previous exposure to OTL38
2. Any medical condition that in the opinion of the investigators could potentially jeopardize the safety of the subject
3. History of anaphylactic reactions to folate, including synthetic folic acid (pteroylmonoglutamic acid) and contrast agents containing indocyanine green for near infrared imaging. Subjects with a medical history of 'idiopathic anaphylaxis' will require evaluation.
4. History of allergy to any of the components of OTL38, including folic acid
5. A positive serum pregnancy test at Screening or a positive urine pregnancy test on the day of surgery or day of admission for female subjects of childbearing potential
6. Clinically significant abnormalities on electrocardiogram (ECG) at screening.
7. Presence of any psychological, familial, sociological condition or geographical challenges potentially hampering compliance with the study protocol and follow-up schedule
8. Impaired renal function defined as eGFR< 50 mL/min/1.73m2
9. Impaired liver function defined as values > 3x the upper limit of normal (ULN) for alanine aminotransferase (ALT) or aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >2x ULN for total bilirubin except in subjects with Gilbert's syndrome.
10. Received an investigational agent in another investigational drug or vaccine trial within 30 days prior to the administration of study drug
11. Known sensitivity to fluorescent light

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, MD, Principal Investigator — University of Pennsylvania
Locations (12):
- United States (12):
  - Stamford, Stamford, Connecticut
  - University of Iowa, Iowa City, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Swedish Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject dosed and withdrawal by subject prior to surgery
Period: Overall Study
Arm/Group | Near-Infrared Imaging Group | No Imaging Group
Started | 100 | 12
Completed | 100 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Near-Infrared Imaging Group | No Imaging Group | Total
Number analyzed (Participants) | 100 | 11 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 5 | 41
  >=65 years | 64 | 6 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9.68) | 64 (9.88) | 65.9 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 9 | 70
  Male | 39 | 2 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 99 | 11 | 110
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 88 | 8 | 96
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 100 | 11 | 111

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Events (CSE)
Description: The primary efficacy endpoint is the proportion of patients who demonstrate at least one CSE as a result of utilizing OTL-38 and Near Infrared Imaging.
Time Frame: 1 day
Population: Full Analysis Set (FAS): The FAS for the primary analysis of the primary efficacy endpoint will include subjects exposed to OTL38 and randomized to undergo fluorescent imaging (OTL38+Imaging) who:
  • Were evaluated under both normal light/palpation and NIR fluorescent light imaging
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Full Analysis Set (FAS): The full analysis set will include subjects exposed to OTL38 and randomized to undergo NIR fluorescent imaging (OTL38+Imaging) who were evaluated under both normal light and NIR fluorescent light imaging
Arm/Group | Full Analysis Set (FAS)
Number analyzed (Participants) | 100
proportion of participants | .530 [.428 to .631]

2. Primary Outcome: Localization of Primary Nodule
Description: Proportion of FAS subjects with one or more primary NIR fluorescence positive lung nodules (cancerous or non-cancerous, excluding normal lung parenchyma) not detected under normal light and/or palpation
Time Frame: 1 day
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Fully Analysis Set (FAS): The full analysis set will include subjects exposed to OTL38 and randomized to undergo NIR fluorescent imaging (OTL38+Imaging) who were evaluated under both normal light and NIR fluorescent light imaging
Arm/Group | Fully Analysis Set (FAS)
Number analyzed (Participants) | 100
proportion of participants | .190 [.118 to .281]

3. Primary Outcome: Identification of Cancerous Synchronous Lesions
Description: The proportion of FAS subjects with one or more NIR fluorescence positive cancerous synchronous lesions not detected under normal light and/or palpation
Time Frame: 1 day
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Fully Analysis Set (FAS)
Number analyzed (Participants) | 100
proportion of participants | .080 [.035 to .152]

4. Primary Outcome: Positive Resection Margins
Description: The proportion of FAS subjects with the identification of a cancerous positive margin that fluoresces within (less than or equal to) 10 mm of the surgical resection staple line
Time Frame: 1 day
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Fully Analysis Set (FAS)
Number analyzed (Participants) | 100
proportion of participants | .380 [.285 to .483]

5. Secondary Outcome: Sensitivity for Cancerous Primary Nodules and Synchronous Lesions in FAS Subjects
Description: Sensitivity or True Positive Rate (TPR) for OTL38 used with fluorescent light in FAS subjects, defined as the proportion of fluorescent light positive primary nodules and synchronous lesions that are histologically confirmed to be cancer relative to the total number of primary nodules and synchronous lesions confirmed to be cancer.
Time Frame: 1 day
Population: Total number of Subjects with Evaluated Tissues
Measure: Number (95% Confidence Interval); unit: proportion of lesions
Units Other Than Participants: Lesions
Arm/Group | Fully Analysis Set (FAS)
Number analyzed (Participants) | 89
Number analyzed (Lesions) | 104
proportion of lesions | .765 [.667 to .842]

6. Secondary Outcome: False Positive Rate for Cancerous Primary Nodules and Synchronous Lesions in FAS Subjects
Description: False Positive Rate (FPR) for OTL38 used with fluorescent light in FAS subjects, defined as the proportion of fluorescent light positive primary nodules and synchronous lesions that are histologically confirmed not to be cancer relative to the total number of fluorescent light positive primary nodules and synchronous lesions
Time Frame: 1 day
Population: Total number of Subjects with Evaluated Tissues
Measure: Number (95% Confidence Interval); unit: proportion of lesions
Units Other Than Participants: Lesions
Arm/Group | Fully Analysis Set (FAS)
Number analyzed (Participants) | 78
Number analyzed (Lesions) | 108
proportion of lesions | .258 [.182 to .352]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of screening through 28 days (+/- 4 days) post-study drug administration
Arm/Group | Near-Infrared Imaging Group | No Imaging Group
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/11
Serious Adverse Events (participants affected / at risk) | 7/100 | 2/11
Other Adverse Events (participants affected / at risk) | 98/100 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Near-Infrared Imaging Group (N=100) | No Imaging Group (N=11)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatic haematoma (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Near-Infrared Imaging Group (N=100) | No Imaging Group (N=11)
Procedural pain (Injury, poisoning and procedural complications) | 78 (88) | 10 (12)
Incision site pain (Injury, poisoning and procedural complications) | 13 (26) | 1 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 28 (29) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 0 (0)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 21 (26) | 1 (2)
Constipation (Gastrointestinal disorders) | 17 (17) | 2 (2)
Hypertension (Vascular disorders) | 11 (15) | 2 (2)
Hypotension (Vascular disorders) | 8 (8) | 1 (1)
Fatigue (General disorders) | 7 (7) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
Urinary retention (Renal and urinary disorders) | 7 (8) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT04241315/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT04241315/SAP_001.pdf